CLINICAL TRIAL: NCT01214122
Title: A Phase I, Open Label, Fixed Sequence, Single Centre Study in Healthy Volunteers to Investigate the Effects of Repeated Oral Doses AZD9668 on the Pharmacokinetics and Pharmacodynamics of a Single Dose of Warfarin
Brief Title: A Drug-Drug Interaction Study Between AZD9668 and Warfarin to Study the Effect of AZD9668 on the Metabolism and Effect of Warfarin
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Masking: None | Purpose: Basic Science
Other Study IDs: D0520C00013; 2010-022360-12 (EudraCT Number)
Record Dates: First submitted 2010-09-21; First posted 2010-10-04 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Pharmacokinetics; Pharmacodynamics
Keywords: Phase 1; Drug-Drug interaction; warfarin; AZD9668; resulting from AZD9668 and Warfarin interaction; pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): AZD9668 - 2 x30mg tablets
  Interventions: Drug: AZD9668
- Treatment B (Experimental): Warfarin - 10 x2.5 mg tablets
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: AZD9668 — 60 mg orally twice daily for 11 days
  Arms: Treatment A
Drug: Warfarin — 10 x 2.5 (25) mg orally once daily on day 1 and on day 14
  Arms: Treatment B

SUMMARY:
The primary purpose of this study is to determine whether the treatment with AZD9668 will affect the metabolism and effect of Warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent (including genotyping screening sample for CYP2C9 and VKORC1) prior to any study specific procedures
* Subjects must be willing to use a barrier method of contraception, unless their partners are post-menopausal or surgically sterile, or if a female partner is of childbearing potential the subject must use a barrier method of contraception (condom) and the partner must use accepted contraceptive methods (oral contraceptive, implant, long term injectable contraceptive or intrauterine device), from first dose of IP (warfarin and AZD9668) until 3 months after last dose of IP (warfarin and AZD9668)
* Have a body mass index between 19 and 30 kg/m2 (inclusive) and a weight between 50 and 100 kg (inclusive)
* Be a non-smoker or ex-smoker who has stopped smoking for >6 months prior to Visit 1.

Exclusion Criteria:

* Any clinically significant disease or disorder
* Subject predicted to have high sensitivity to warfarin based on CYP2C9 and VKORC1 genotypes
* Any clinically relevant abnormal findings in physical examination

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 1
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 2
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 3
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 4
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 5
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 6
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 7
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 8
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 9
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 10
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 11
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 12
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 13
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 14
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 15
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 16
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 17
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 18
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 19
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 20
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 21
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 22
Pharmacokinetics for (R)- and (S)- Warfarin, measured by maximum plasma concentration (Cmax ) and area under the plasma concentration-time curve (AUC) | Pharmacokinetic (PK) sampling will be performed day 23
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 1
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 2
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 3
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 4
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 5
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 6
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 7
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 8
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 9
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 10
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 11
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 12
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 13
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 14
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 15
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 16
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 17
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 18
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 19
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 20
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 21
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 22
Pharmacodynamics measured by maximum international normalised ratio ( INRmax) | International normalised ratio (INR) sampling will be performed day 23

SECONDARY OUTCOMES:
Pharmacokinetics for AZD9668 measured by Css,max | Range from day 9 to 23
Pharmacokinetics for AZD9668 measured by tss,max | Range from day 9 to 23
Pharmacokinetics for AZD9668 measured by Css,min | Range from day 9 to 23
Pharmacokinetics for AZD9668 measured by CLss/F | Range from day 9 to 23
Severity of Adverse Events as a Measure of Safety and Tolerability | Adverse events will be collected pre-dose, during treatment and at follow up
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Adverse events will be collected pre-dose, during treatment and at follow up
Pharmacokinetics for (R)- and (S)- Warfarin measured tmax. | Range from day 1 to 23
Pharmacokinetics for (R)- and (S)- Warfarin measured t½. | Range from day 1 to 23
Pharmacokinetics for (R)- and (S)- Warfarin measured CL/F. | Range from day 1 to 23
Pharmacokinetics for (R)- and (S)- Warfarin measured Vz/F. | Range from day 1 to 23

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D O'Brien, MD, PhD, Study Director — AstraZeneca R&D; Ingemar Bylesjö, MD, Principal Investigator — Berzelius Clinical Reseach Centre; Wolfgang Kühn, MD, Principal Investigator — Quintiles AB, Phase 1 Services
Locations (2):
- Sweden (2):
  - Research Site, Linköping
  - Research Site, Uppsala